CLINICAL TRIAL: NCT04288843
Title: Endometrial Dating by Ex-vivo Imaging of Endometrial Biopsies of In-vitro Fertilization Candidate Participants
Status: Completed | Type: Observational
Sponsor: Fertigo Medical Ltd (Industry)
Collaborators: Kaplan Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: FER-CT-001
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2022-03

CONDITIONS: Endometrium
Keywords: Endometrial dating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Pipelle biopsy of the endometrium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the correlation between cycle day determination by clinical signs, study participant testimony, endometrium histopathology biopsy and ex-vivo imaging of the uterus endometrium.

DETAILED DESCRIPTION:
In order to assess the efficacy of using ex-vivo endometrial imaging to determine optimal time for embryo transfer, two to four separate analyses, including imaging, and the current standard method of endometrial dating (ultrasound, histological and blood tests) will be performed as well as participant's testimony. Dating by hormonal profile (blood tests) will be contingent on availability of the tests for each subject. So shall be the ultrasound test. During the analysis data will be acquired for subsequent correlation analysis. In addition, a parallel in-vivo analysis, similar in methodology to the ex-vivo analysis, may be performed via imaging by hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Female
2. Age: 18-40
3. Belong to one of the three following groups:

   1. Women undergoing fertility treatment, and are regularly ovulating
   2. Women whose fertility status is unknown
   3. Women proved to be fertile (previous spontaneous successful pregnancy)

Exclusion Criteria:

1. Women with known existing endometrial pathology
2. Women with known history of infertility due to oligo-ovulation or anovulation.
3. Women with medical history of malignant tumors in their reproductive system
4. Women that are on any hormonal medications or treatments (excluding hormonal contraception in previous cycles)
5. Women that are on hormonal contraception treatment in their current cycle
6. Women with intrauterine device
7. Women menstruating on the day of the biopsy collection

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females
Study Population: The study will include up to 200 women between the ages of 18 - 40, to be recruited from the general population and medical center patient population, after determination that they are suited to the study according to the inclusion/exclusion criteria, and after having given informed consent to participate in the study.
  The sample size of the study will be determined such that adequate mapping of the 24 days of the menstrual cycle (putting more weight on luteal phase), excluding menstruation days (assuming a 28 day cycle), and dividing of the cohort into subgroups by age, can be achieved using the study methods described below, while adhering to financial constraints.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-06-16 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Correlation between image-based endometrial dating and that of histology | 12 months
  Correlation coefficients and/or P-value levels

SECONDARY OUTCOMES:
Correlation between image-based endometrial dating and other collected data | 12 months
  Collected data: hormonal profile, ultrasound images, subject self-reporting of cycle date

CONTACTS AND LOCATIONS:
Overall Officials: Tsafrir S Kolatt, Ph.D., Study Chair — Fertigo Medical Ltd
Locations (2):
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot

IPD SHARING:
Plan to Share IPD: Undecided